CLINICAL TRIAL: NCT05421702
Title: Surgical, Pathological and Oncological Outcomes of Laparoscopic Conventional Colectomy Versus Complete Mesocolic Excision for Operable Colon Cancer Cases in Upper Egypt
Brief Title: Comparison Between Results of 2 Laparoscopic Surgical Procedures in Operable Colon Cancer Cases in Upper Egypt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mostafa Farrag Mohammed, assistant lecturer of general surgery, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-06-17
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Colon Cancer Stage I; Colon Cancer Stage II
Keywords: Colon cancer; Colectomy; Mesocolic; Conventional; Laparoscopic; Surgical; Pathological
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Operable colon cancer cases
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Operable colon cancer cases (Active Comparator): All patients with operable colon cancer who will undergo laparoscopic conventional colectomy
  Interventions: Procedure: laparoscopic conventional colectomy
- Group B Operable colon cancer cases (Active Comparator): All patients with operable colon cancer who will undergo laparoscopic complete mesocolic excision
  Interventions: Procedure: laparoscopic complete mesocolic excision

INTERVENTIONS:
Procedure: laparoscopic conventional colectomy — Laparoscopic colectomy with only lymph node dissection up to level 2 lymph nodes D2.
  Other Names: D2 colectomy
  Arms: Group A Operable colon cancer cases
Procedure: laparoscopic complete mesocolic excision — Laparoscopic colectomy with lymphovascular dissection from level 3 lymph nodes or more D3.
  Arms: Group B Operable colon cancer cases

SUMMARY:
The investigators will assess and compare Surgical, pathological and oncological outcomes between two laparoscopic procedures conventional colectomy versus complete mesocolic excision for operable colon cancer cases in Upper Egypt

DETAILED DESCRIPTION:
Colon cancer is considered a huge clinical surgical burden accounting for 10% of cancer cases and deaths all over the world with consideration that surgery and adjuvant chemotherapy(if indicated) are the main lines of treatment .

When Werner Hohenberger and colleagues described complete mesocolic excision (CME) in 2009; resection along the embryological and lymphovascular planes with appropriate resection margins, they did it for years before describing it with suggestion of improved disease outcomes and overall survival compared to the conventional colectomy (CC).

The principles of CME were described after the significant improvement of rectal adenocarcinoma surgical outcomes with establishment of total mesorectal excision (TME) in which tumor resection is associated with dissection of mesorectal fascial embryologic and lymphovascular planes.

CME includes the same principles of the CC with maximizing lymph node dissection level into (D3 extended lymphadenectomy instead of D1 and D2 in conventional colectomy) and central vascular ligation (CVL) of the main feeding vessel(s) at their origin, with suggested improved disease-free and overall survival with suggested superior pathological and oncological results in the specimen.

Some surgeons consider that CME; with D3 extended lymphadenectomy and CVL is the optimal or standard surgical method in primary cancer colon based on suggested reduced local recurrence and improved disease-free and overall survival.

Although CME has a theoretical advantages and promising early results, it is not widely adopted as the standard in some areas. CME is technically more demanding than CC and suggested to be associated with more intraoperative visceral injuries and non-surgical complications and many doubts persist about safety and efficacy of the procedure.

The questions of interest and research, should CME be regarded as the optimal procedure for colon cancer cases? And also another question; is conventional colectomy suboptimal?

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes will be included.
2. Age: all adult patients.
3. All diagnosed patients with operable cancer colon.
4. Cancer at cecum, appendix, ascending colon, hepatic flexure or at splenic flexure, transverse and descending colon and sigmoid colon.
5. Fit patients.

Exclusion Criteria:

1. Irresectable colon cancer.
2. Inoperable colon cancer.
3. Rectal cancer.
4. Unfit patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-07-21 (Actual)

PRIMARY OUTCOMES:
Postoperative lymph node status | 2 weeks postoperative
  Histopathological examination of the resected colon with lymph node status and number
Postoperative histopathological result | 2 weeks postoperative
  Type of the colon cancer
Occurence of anastomotic leak | within 4 weeks postoperative
  Yes/No
Amount of anastomotic leak | within 4 weeks postoperative
  Amount in cubic cm and nature of it with its management
Intraoperative visceral injury type | Intraoperative reporting
  Yes/No and its type
Intraoperative visceral injury management | Intraoperative reporting
  How managed
Postoperative complications | 4 weeks postoperative
  Yes/No with Reporting the postoperative complications; according to the Clavien-Dindo Grading System
Operative time | Reporting immediately postoperative (at end of operation)
  Reporting operative time with measurements in minutes
Intraoperative vascular injury | Intraoperative
  Yes/No with measurement in Cubic Cm and how managed
Intraoperative blood loss | Intraoperative
  Yes/No with measurement in Cubic Cm
Resection margins in postoperative histopathological status | 2 weeks postoperative
  Free or invaded
Postoperative peritonitis | 4 weeks postoperative
  Cause and how to manage?
Colon cancer stage | 2 weeks Preoperative
  According to primary tumor, regional nodes, metastasis (TNM) staging system
Postoperative faecal fistula | 12 weeks postoperative
  Reporting Yes/No with amount in cm3 and management
length of resected mesocolon | 2 weeks postoperative
  In cm
Urological complications | Intraoperative and 4 weeks postoperative
  Type and management
Carcinoembryonic antigen (CEA) level | 2 weeks preoperative
  Carcinoembryonic antigen (CEA) level by ng/mL
Type of anastomosis | Intraoperative
  Type of anastomosis (intra- or extracorporeal)

SECONDARY OUTCOMES:
Age | preoperative
  In years
Preoperative haemoglobin level | preoperative
  measured by g/dl
Type of colonic anastomosis | Intraoperative
  Stapler or hand sewing
Preoperative histopathological result | 2 weeks preoperative
  Histopathological examination
Neoadjuvant therapy | 2 weeks Preoperative
  Type of the neoadjuvant and duration
Site of cancer colon | 2 weeks preoperative
  cecum, appendix, ascending colon, hepatic flexure or at splenic flexure, transverse and descending colon and sigmoid colon
Neurological complications | 4 weeks postoperative
  Type and management
Preoperative preparation | 3 days Preoperative
  Mechanical and/or chemical
Cardiopulmonary complications | 4 weeks postoperative
  Yes/No Cardiopulmonary complications type and how managed
Conversion to open surgery | intraoperative
  Yes/No with the cause
application of subcutaneous suction | 1 week Postoperative
  Yes/No
Average daily amount in subcutaneous suction | 2 weeks Postoperative
  in Milliliters
Average daily amount in intraperitoneal drain | 2 weeks Postoperative
  in Milliliters
Wound infection | 2 weeks postoperative
  Yes/No and how managed
Postoperative ileus | 2 weeks postoperative
  Postoperative ileus Yes/No
Hospital stay | 4 weeks postoperative
  In days
Wound dehiscence | 4 weeks postoperative
  Yes/No
Preoperative colonoscopic examination result | 2 weeks preoperative
  mass/ulcer

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed E Ahmed, Professor, Study Chair — Sohag University; Mena Z Helmy, Ass prof., Study Director — Sohag University; Mostafa F Mohammed, Ass lecturer, Principal Investigator — Sohag University
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available.